CLINICAL TRIAL: NCT02401724
Title: A Randomised Trial of Non-Invasive Brain Stimulation (NIBS) in Stroke Survivors
Brief Title: NonInvasive Brain Stimulation in Stroke Patients
Acronym: RTNIBS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GN13NE562
Record Dates: First submitted 2015-03-10; First posted 2015-03-30 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2015-03

CONDITIONS: Stroke
Keywords: Hemispatial neglect; Transcranial direct current stimulation; Rehabilitation
MeSH Terms: conditions — Stroke; Perceptual Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Action Training (Active Comparator): Training exercise which involves patients lifting up rods of different sizes and shifting their grip if this is too far to one side
  Interventions: Other: Action Training
- tDCS (Experimental): A constant 1mA current will be applied to the left (undamaged) side of the scalp with an electrode covered with a damp cotton pad (25 cm2). The current will be applied for 15 minutes per day, with a total of 10 sessions over 3 weeks.
  Interventions: Other: Transcranial direct current stimulation
- Action Training + tDCs (Experimental): This will involve the same procedure as in action training only but with tDCS applied for 15 minutes during the rodlifting.
  Interventions: Other: Transcranial direct current stimulation; Other: Action Training
- Control training (Placebo Comparator): For the control training, patients will be asked to simply reach for the right hand side of each rod with their right (unaffected) hand and lift it

INTERVENTIONS:
Other: Transcranial direct current stimulation
  Other Names: tDCS
  Arms: Action Training + tDCs; tDCS
Other: Action Training
  Arms: Action Training; Action Training + tDCs

SUMMARY:
After a stroke affecting the right side of the brain, many patients are affected by "spatial neglect": the damage to the brain causes them to ignore the left side of their surroundings. At its most extreme they may be unaware that they have a left side, or believe that it is moving normally when it is in fact paralysed. In milder cases, people may be unable to recognise touch on the left side if their right side is also being touched, or objects in their left visual field if something is visible to their right. Neglect alters peoples' quality of life profoundly, often renders them more dependent on others to undertake basic activities of daily living, and makes effective rehabilitation much more difficult.

The limited success of current treatment approaches indicates gaps in understanding of the underlying mechanisms of neglect and its recovery. Recent data suggest that the problems in responding to the left side are a result of an imbalance of activity in those parts of the brain responsible for deciding which side to pay attention to. It might therefore be possible to help people with neglect by "rebalancing" the brain either by increasing activity in the damaged side, or alternatively by reducing activity in the undamaged side. In this pilot study, the investigators will test whether they can help by doing the second of these things.

The investigators propose to conduct a pilot clinical trial to explore whether using electric currents to temporarily modify the activity of specific areas of the intact side of the brain, influences recovery from neglect, when used either alone, or in combination with a training method that has previously appeared promising as a treatment. Brain activity will be modified using a technique called "transcranial direct current stimulation (tDCS)", in which small electric currents are applied to the scalp with a wire covered in damp cotton pads. This will be done over the specific parts of the brain that are responsible for focusing attention to one side.

The investigators will compare the clinical outcomes of four interventions (1: behavioural, 2: tDCS, 3: a combination of both and 4: control).

The investigators hope that these studies will advance their understanding of what treatments may help people with neglect, and how they might work.

ELIGIBILITY:
Inclusion Criteria:

1. Ischemic stroke affecting the right hemisphere, confirmed by CT or MRI.
2. Persistent neglect for one month after ictus (confirmed by BIT).
3. Prestroke functional independence (modified Rankin Scale score 0-2).
4. Between 18-90 years of age

Exclusion Criteria:

1. Patients younger than 18.
2. Patients who do not understand verbal or written English (ie.need of translaters)
3. bilateral infarcts (Confirmed by CT, MRI)
4. Dementia (MOCA, Score <26).
5. Neurological Disease (eg. Parkinson's Disease, epilepsy, MS)
6. Significant morbidity (eg cancer, severe cardiac failure) likely to affect participation.
7. Alcohol excess (more than 50/40 units a week for men/women respectively).
8. Patients who fall under the exclusion criteria for TDCS which includes patients suffering from a stroke related seizure :

History of epilepsy, medications or psychoactive drugs that can lower seizure threshold [imipramine, amitriptyline, doxepine, nortriptyline, maprotiline, chlorpromazine, clozapine, foscarnet, ganciclovir, ritonavir, amphetamines, cocaine, (MDMA, ecstasy), phencyclidine (PCP, angel dust), ketamine, gammahydroxybutyrate (GHB), alcohol, theophylline]. Withdrawal from alcohol, barbiturates, benzodiazepines, meprobamate, chloral hydrate. Patients who are pregnant or have suffered from a stroke-related seizure.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-03; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Change in Behavioural Inattention Test (BIT) | 6 months post intervention

SECONDARY OUTCOMES:
Compliance as measured by adherence to task instructions (percentage of intervention sessions, BIT tests completed) | baseline
Compliance as measured by adherence to task instructions (percentage of intervention sessions, BIT tests completed) | 3 weeks
Compliance as measured by adherence to task instructions (percentage of intervention sessions, BIT tests completed) | 6 months
Retention Numbers | baseline
Retention Numbers | 3 weeks
Retention Numbers | 6 months

REFERENCES:
- [Derived] Longley V, Hazelton C, Heal C, Pollock A, Woodward-Nutt K, Mitchell C, Pobric G, Vail A, Bowen A. Non-pharmacological interventions for spatial neglect or inattention following stroke and other non-progressive brain injury. Cochrane Database Syst Rev. 2021 Jul 1;7(7):CD003586. doi: 10.1002/14651858.CD003586.pub4. PMID 34196963
- [Derived] Elsner B, Kugler J, Pohl M, Mehrholz J. Transcranial direct current stimulation (tDCS) for improving activities of daily living, and physical and cognitive functioning, in people after stroke. Cochrane Database Syst Rev. 2020 Nov 11;11(11):CD009645. doi: 10.1002/14651858.CD009645.pub4. PMID 33175411
- [Derived] Learmonth G, Benwell CSY, Marker G, Dascalu D, Checketts M, Santosh C, Barber M, Walters M, Muir KW, Harvey M. Non-invasive brain stimulation in Stroke patients (NIBS): A prospective randomized open blinded end-point (PROBE) feasibility trial using transcranial direct current stimulation (tDCS) in post-stroke hemispatial neglect. Neuropsychol Rehabil. 2021 Sep;31(8):1163-1189. doi: 10.1080/09602011.2020.1767161. Epub 2020 Jun 5. PMID 32498606